CLINICAL TRIAL: NCT07116590
Title: Investigation of Cervical Spinal Stability, Proprioception, and Body Awareness in Individuals With Migraine
Brief Title: Cervical Stability and Body Awareness in Migraine
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Güngör Beyza ÖZVAR, Principal Investigator, Hacettepe University
Other Study IDs: Migraine
Record Dates: First submitted 2025-08-06; First posted 2025-08-11 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Migraine
Keywords: migraine; body awareness; cervical spinal stability; cervical proprioception
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Migraine: Patients diagnosed with migraine without aura according to the International Classification of Headache Disorders (ICHD-III) criteria, currently in the interictal period, aged between 18 and 55 years, and who agree to participate in the study will be included.
- Healthy subjects: Individuals matched with the migraine group in terms of age and sex distribution.

SUMMARY:
The aim of this study is to compare cervical spinal stability, cervical proprioception, and body awareness in individuals with migraine and healthy controls, and to examine the relationship between these parameters.

Hypotheses of the Study:

H1: Cervical spinal stability differs between individuals with migraine and healthy individuals.

H2: Cervical proprioception differs between individuals with migraine and healthy individuals.

H3: Body awareness differs between individuals with migraine and healthy individuals.

H4: There is a relationship between cervical spinal stability, cervical proprioception, and body awareness in individuals with migraine.

DETAILED DESCRIPTION:
After collecting demographic and disease-related data from individuals with migraine, and demographic data from healthy controls, the following assessments will be conducted: Migraine Disability Assessment Questionnaire (MIDAS), Bournemouth Neck Questionnaire, Fremantle Neck Awareness Questionnaire, Body Awareness Questionnaire, Body Awareness Rating Questionnaire, cervical spinal stability, and cervical proprioception.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with migraine without aura according to the International Classification of Headache Disorders (ICHD-III) criteria,
* Are in the interictal period,
* Are between 18 and 55 years of age, and
* Agree to participate in the study

  * Age- and sex-matched healthy individuals

Exclusion Criteria:

* Individuals with other types of headache,
* Those with a history of neck or head trauma,
* Individuals with cervical disc herniation or cervical arthrosis,
* Those with any other systemic or neurological medical condition (e.g., chronic pain syndrome, rheumatoid arthritis, systemic lupus erythematosus, stroke, trigeminal neuralgia, etc.),
* Pregnant individuals,
* Patients who have received anesthetic blockade within the past 6 months.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: migraine patients and healthy subjects with inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Migraine Disability Assessment Questionnaire-MIDAS | up to 3 months
  It is a questionnaire consisting of five questions related to disability over the past three months. Individuals score the number of days lost due to headache in three domains: schoolwork, paid work, and household activities. Additionally, they report the number of extra days with significant activity limitations (defined as at least a 50% reduction in productivity) in paid and household work. The MIDAS score is calculated by summing the scores of these five items.
Bournemouth Neck Questionnaire: | up to 3 months
  This questionnaire consists of seven items, each scored on a scale from 0 to 10. It evaluates the impact of pain on daily activities, pain severity, levels of anxiety and depression, kinesiophobia, and the ability to cope with pain.
Fremantle Neck Awareness Questionnaire | up to 3 months
  This questionnaire consists of nine items, each scored on a scale from 0 to 4. It assesses awareness of the cervical region. Higher scores indicate poorer body awareness.
Body Awareness Questionnaire | up to 3 months
  This questionnaire consists of 18 items, each scored on a scale from 1 to 7, and is used to assess body awareness. Higher scores indicate better body awareness.
Body Awareness Rating Questionnaire | up to 3 months
  This questionnaire consists of 24 items divided into four domains: function, mood, sensation/emotion, and awareness. Each item scores a 7-point Likert type scale. Each factor's scores range between 6 to 42 and higher scores indicates higher body awareness
Cervical Spine Stability | up to 3 months
  The craniocervical flexion test will be performed using a pressure biofeedback unit (Stabilizer, Chattanooga, Australia). The test consists of five stages. During the test, participants will lie in a supine position with the head and neck in neutral alignment, and the device will be placed under the suboccipital region.
  In the initial stage, the pressure will be set at 20 mmHg, and participants will be instructed to perform a craniocervical flexion movement. Subsequently, the test will proceed through five incremental stages, increasing the pressure in 2 mmHg increments from the initial 20 mmHg up to a maximum of 30 mmHg.
  At each pressure level, participants will be asked to maintain the movement for 10 repetitions of 10 seconds each. Based on these stages, the Activation Score and Performance Index will be calculated
Cervical Proprioception | up to 3 months
  Joint position error test will be conducted using a laser pointer attached to the participant's head. While sitting on a chair with back support, participants will face a wall where a target will be placed 90 cm away.
  Participants will first be asked to sense the starting position (the center of the target). Then, with their eyes closed, they will be instructed to return their head to the starting position from various directions (flexion, extension, and rotation).
  The deviation from the target center will be measured in centimeters, and the test will be repeated three times. The average of the three trials will be used as the final score.

CONTACTS AND LOCATIONS:
Overall Officials: Esranur Özoğul, Principal Investigator — Yuksek Ihtisas University; Büşra Kalkan Balak, Principal Investigator — Yuksek Ihtisas University
Locations (1):
- Yuksek Ihtisas University, Ankara, Balgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No